CLINICAL TRIAL: NCT04117438
Title: Interviewing Breast Cancer Patients to Understand the Patients Relationship With Food Before and After Cancer Diagnosis.
Brief Title: Tell us Your Food Story
Status: Withdrawn | Type: Observational
Why Stopped: Due to COVID-19 pandemic, we will not be pursuing this study
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Amy Rymaszewski, Research Associate II, Medical College of Wisconsin
Other Study IDs: PRO00034502
Record Dates: First submitted 2019-10-02; First posted 2019-10-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — There is no intervention. We are just asking breast cancer patients what their food story is.

SUMMARY:
In 2017, it is estimated that 318,590 Americans, men and women, will be diagnosed with breast cancer (American Cancer Society, 13). It was predicted in the 1970s that 1 in 11 Americans would be diagnosed with breast cancer, currently, it is 1 in 8 people. A person is twice as likely to be diagnosed with breast cancer if they have one first-degree female with a diagnosis, 3-4 times if there is more than one first-degree female relative with a diagnosis. Reasons for this increase in breast cancer diagnoses are that people are living longer, changes in reproductive patterns, increases or decreases in menopausal hormone use, increased numbers of detection through screening including genetic testing, and the rising prevalence of obesity (American Cancer Society). The purpose of this study is to better understand how a diagnosis of breast cancer supports change in diet and their food story.

Qualitative methodology and specifically the long interview is the method the team will use to gain insight into adult patients' perceptions of their food story.

DETAILED DESCRIPTION:
1. All interviews will occur at a community clinic or convenient community location.
2. Clinical faculty will receive an oral and written overview of the project prior to beginning in case they have patients they want to recommend to participate.
3. Physician will approach individual patients to participate during a regular medical office visit, patients will be given an introduction and overview of the study, and then will be asked if they would like to participate in the study.
4. If the patient wants to participate, Malika Siker, MD will schedule a time for the patient to meet with a member of the study team to conduct the interview.
5. The interview will be scheduled at a time convenient for the patient.
6. If the patient does not want to participate, no further action is required
7. All study subjects will be adults with the ability to understand the study and consent to participate.
8. The sample will be a convenience sample based upon interest in participating.
9. At the time of the interview, patients will receive a written and oral overview of the research.
10. The subject will have ample time to ask questions before completing the survey or beginning the interview.

    All study subjects will understand and agree to having the interview audiotaped.
11. The interview will take place immediately after the subject has agreed to participate.
12. Interviews will last between approximately 60 minutes. Subjects can decline to answer any question and can withdraw from the study at any time during the process.
13. Our highest estimate is that 50 subjects will be needed to complete the project.
14. Interviews will be audiotaped and transcribed verbatim by a transcription service following the conclusion of the interview.
15. The transcriptionist will be instructed to remove any names of individuals that may be discussed by the subject.
16. Transcriptions will be placed in a password protected computer file.
17. PI will review the transcripts to ensure that transcriptions are anonymous.
18. When determined, PI will instruct that the recording be erased.
19. The team will only begin analysis after ensuring that all transcripts are anonymous.
20. The team will analyze the data for thick description and for themes that emerge during the analysis by following procedures developed by Corbin and Strauss.

ELIGIBILITY:
Inclusion Criteria:

* Any patient that lives in Southeastern Wisconsin and has a diagnosis of breast cancer, or a history of breast cancer and is over the age of 18.

Exclusion Criteria:

* Any subject that is under the age of 18, that does not live in Southeastern Wisconsin and has no diagnosis of breast cancer, or a history of breast cancer will be excluded.

Max Age: 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Little is known about a patient and their food stories before, during and after cancer treatment. The investigators would like to understand how cancer impacts a patients food narrative. Patients that live in areas where food is less readily accessible maybe looking for ways to improve their food narrative. This population will only include any 18 or older adult with a history of breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Breast cancer patients relationship with food. | 10 years
  A patient recently diagnosed with breast cancer will be more aware of the relationship they have with diet then those patients that have been in treatment for an extended period of time. The investigators will analyze the data for thick description and for themes that emerge during the analysis by following procedures developed by Corbin and Strauss.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Since these are personal stories, the investigators will not be sharing these with others.